CLINICAL TRIAL: NCT06650904
Title: The Effect of Simulation-Based Child and Family Communication Practice on Pediatric Nurses' Communication and Problem-Solving Skills
Brief Title: Simulation Based Child and Family Communication Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ebru Kilicarslan Toruner, Nursing Faculty, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021 - 1039
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Nursing; Communication; Problem Solving
Keywords: pediatric nursing; communication; problem-solving; simulation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: 48 nurses serving pediatric patients working in a private hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation-Based Child and Family Communication Application (Other): pre-test post-test design quasi-experimental study without control group
  Interventions: Other: simulation based training

INTERVENTIONS:
Other: simulation based training — Simulation practice enables the acquisition of realistic skills. Semi-structured scenarios used in the training allow nurses to demonstrate their real communication skills.

SUMMARY:
The use of simulation-based methods in training pediatric nurses plays an important role in improving their communication skills. In this context, the aim of the research is to develop a simulation-based child and family communication training program. The study aims to evaluate the effect of this communication practice on the communication and problem-solving skills of pediatric nurses. The research is designed as a quasi-experimental study. The study sample will consist of 48 nurses working in pediatric clinics. The nurses, who will receive information about the simulation laboratory, will be divided into groups of 3, and the application will be conducted using a semi-structured scenario in the simulation laboratory. The application will be recorded on video, and feedback will be provided through debriefing sessions based on these recordings. A descriptive data form, a simulation self-assessment scale, a communication skills inventory, and an adult problem-solving scale will be used for data collection. Data will be collected before the application, and at the 1st week and 1st month after the application. As a result of the research, it is aimed to adapt the simulation-based communication skills given to pediatric nurses to the clinical environment.

Questions of the study;

Pediatric nurses before and 1 week and 1 month after simulation-based child and family practice:

Is there a difference between the mean scores of the Communication Skills Inventory? Is there a difference between the mean scores of the Problem Solving Inventory?

Pediatric nurses 1 week and 1 month after simulation-based child and family practice:

Is there a difference between the mean scores of the Simulation Self-Assessment Scale?

DETAILED DESCRIPTION:
The research is planned to be conducted as a quasi-experimental study using pre-test-post-test in order to examine the effect of simulation-based applied training for children and families on the communication and problem solving skills of pediatric nurses. The research will be conducted in the pediatric simulation laboratory of Gazi University Faculty of Nursing, Department of Pediatric Nursing. Pediatric Nursing Practice Laboratory consists of two application areas. In the first application area, there is a simulation room and a control room used by the instructors, where student practices are observed and evaluated through mirror glass. The second application area is used to evaluate the analysis phase and feedbacks of the participants' applications, which are videotaped after the simulation applications, by coming together with the participants after the application. The research sample will consist of 48 nurses who work with pediatric patients in a private hospital and agree to participate in the study. After obtaining the necessary permissions for the study, a 4-hour pre-application will be made with a different group of nurses not included in the study and all modules and forms will be applied. The necessary arrangements identified will be made before the application. Simulation application groups will be formed with groups of 3 people on a predetermined day and time according to the working days and hours of the nurses who agree to participate in the study. Before the simulation application, the pediatric simulation laboratory will be introduced to the nurses who agree to participate in the study. The orientation of the nurses to the simulation environment, the materials to be used and the characteristics of the model (expected goal, what they are asked to do, application time, evaluation) will be provided. The pre-created semi-structured scenario for the themes determined before the simulation application will be explained to the nurses. The simulation practice will last approximately 1.5 hours (40 min simulation practice + 50 min debriefing = 1.5 hours). During the implementation, the scenario will be realized with video shooting. While the researchers will manage the scenario, they will take notes on the practices of the nurses. After the simulation application, feedback will be provided to the nurses about the positive aspects and skills that need to be developed by the researchers through a debriefing interview over the video recordings. The data obtained will be evaluated using SPSS 25.0 package program. Data will be evaluated by descriptive analysis (percentage, frequency). The confidence interval will be accepted as 0.95. In the study, firstly, it will be evaluated whether the data obtained show normal distribution or not. Pre-test and post-test scale scores will be analyzed and evaluated with t-test for dependent groups. The cause and effect relationship between the scales will be analyzed by regression analysis. In the analysis of the results, the findings will be considered statistically significant if p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Providing care to a pediatric patient
* Agreeing to participate in the study

Exclusion Criteria:

* Nurses who want to withdraw from the study
* Nurses who have not completed all modules

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Communication Skills Inventory | up to 1 month from the beginning of training
  The inventory used to assess an individual's own communication skills consists of 3 sub-dimensions: mental, emotional and behavioral. The first form, which was used as the "Communication Skills Assessment Scale" developed by Korkut (1996) with 70 items, was revised as the 45-item "Communication Skills Inventory" by Ersanlı and Balcı in 1998 after its validity and reliability was established. The inventory is a 5-point Likert scale. Opposite each statement, there are frequency expressions as "always (5), usually (4), sometimes (3), rarely (2), never (1)". The highest score that can be obtained from the inventory is 225 and the lowest score is 45. The total score obtained from the inventory shows the general communication skill level of the person. In addition, each sub-dimension of the inventory can be evaluated separately. A high score indicates a high level of communication skills. The cronbach alpha reliability coefficient of the scale is 0.72
Problem Solving Inventory | up to 1 month from the beginning of the training
  The scale developed by Heppner and Peterson (1982) is a 6-point Likert-type scale consisting of 35 items that determines the stages of the problem solving process and evaluates what individuals think about their own problem solving behaviors and approaches. The inventory consists of three dimensions: "Solving Problem Confidence", 'Approach-Avoidance Style' and 'Personal Control'. The minimum score of the inventory is 32 and the maximum score is 192. Items 9, 22 and 29 of the inventory are not included in the scoring. The Turkish validity and reliability of the inventory was conducted by Şahin, Şahin, and Heppner (1993). The usability study for nurses was conducted by Erenler (2007). A high score obtained from the inventory indicates that the individual perceives himself/herself as inadequate in problem solving skills. Cronbach alpha internal consistency of the inventory was determined as 0.90.
Self-Assessment Scale for Simulation Laboratory Applications (SES-SLP) | 1 week after the start of training
  The scale developed by Kılıcarslan Toruner et al. (2021) consists of 23 items and 2 sub-dimensions. The sub-dimensions of the scale are developmental factor (19 items) and challenging factor (4 items). The scale is 5-point Likert type. There are five options for each item in the scale: 0 = Disagree, 1 = Somewhat Agree, 2 = Undecided, 3 = Agree and 4 = Strongly Agree. Items 3, 6, 10 and 19 are reverse coded. The minimum score of the scale is 0 and the maximum score is 92. A high score indicates that the individual's perspective on professional knowledge, skills and attitudes has increased due to the practices. The cronbach alpha value of the scale is 0.94

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No